CLINICAL TRIAL: NCT00002226
Title: A Multicenter, Dose Escalating Study in Patients With Cutaneous AIDS-Related Kaposi's Sarcoma
Brief Title: Safety and Effectiveness of Giving SU5416 to HIV-Infected Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SUGEN (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 294A; 5416.003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; Sarcoma, Kaposi; Antineoplastic Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms | interventions — Semaxinib

INTERVENTIONS:
Drug: SU5416

SUMMARY:
The purpose of this study is to see if it is safe and effective to give SU5416 to HIV-infected patients with AIDS-related Kaposi's sarcoma (KS). SU5416 may prevent the growth of KS tumors.

DETAILED DESCRIPTION:
Groups of 3-6 patients are sequentially assigned to receive escalating doses of SU5416 in 33% increments. Study drug is administered as a twice-weekly intravenous injection for 4 weeks. In the absence of unacceptable toxicity, responding patients may continue on SU5416 in 4-week treatment cycles for a maximum of 1 year or until the presence of unacceptable toxicity or tumor progression.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 18 years old.
* Are HIV-positive.
* Have KS with at least 5 skin lesions.
* Have been in stable condition for at least 6 weeks prior to study entry, if receiving antiretroviral therapy.
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have had surgery within 4 weeks of study entry.
* Have taken certain medications, including therapy for KS, within 3 weeks prior to study entry.
* Have pulmonary KS (KS in your lungs).
* Have certain serious medical conditions, including liver or kidney problems, certain infections, and certain cancers.
* Are allergic to Cremophor.
* Have not recovered from previous cancer treatment (chemotherapy, radiotherapy, or immunotherapy).
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Norris Cancer Ctr / USC, Los Angeles, California
  - UCLA Care Ctr / Ctr for Hlth Sciences, Los Angeles, California
  - Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California
  - New York Univ Med Ctr, New York, New York

REFERENCES:
- [Background] Gill P, Arasteh K, Jacobs M, Friedman-Kiel A, Miles S, Gracey S, Hannah A, Langecker P. A multicenter, dose-escalating study in patients with AIDS-related Kaposi's Sarcoma 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29